CLINICAL TRIAL: NCT05132075
Title: A Randomized, Controlled, Open Label, Phase III Study Evaluating the Efficacy and Safety of JDQ443 Versus Docetaxel in Previously Treated Subjects With Locally Advanced or Metastatic KRAS G12C Mutant Non-small Cell Lung Cancer
Brief Title: Study of JDQ443 in Comparison With Docetaxel in Participants With Locally Advanced or Metastatic KRAS G12C Mutant Non-small Cell Lung Cancer
Acronym: KontRASt-02
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJDQ443B12301; 2023-510082-10-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Non small cell lung cancer; Lung cancer; Cancer of the lung; Cancer of lung; Pulmonary Cancer; Neoplasms, Lung; Neoplasms, Pulmonary
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — JDQ443; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JDQ443 (Experimental): Participants will be treated with JDQ443
  Interventions: Drug: JDQ443
- Docetaxel (Active Comparator): Participant will be treated with docetaxel following local guidelines as per standard of care and product labels
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: JDQ443 — JDQ443 tablets, orally administered
  Arms: JDQ443
Drug: docetaxel — docetaxel concentrated solution for infusion, intravenously administered
  Arms: Docetaxel

SUMMARY:
This is a phase III randomized open label study designed to compare JDQ443 as monotherapy to docetaxel in participants with advanced non-small cell lung cancer (NSCLC) harboring a KRAS G12C mutation who have been previously treated with a platinum-based chemotherapy and immune checkpoint inhibitor therapy either in sequence or in combination.

DETAILED DESCRIPTION:
The study has been designed as a Phase III trial and consists of 2 parts:

* Randomized part will evaluate the efficacy and safety of JDQ443 as monotherapy in comparison with docetaxel. Participants randomized to docetaxel arm will have the opportunity to cross-over to JDQ443 at disease progression per RECIST 1.1 confirmed by BIRC.
* Extension part will be open after final progression-free survival (PFS) analysis (if the primary endpoint has met statistical significance) to allow participants randomized to docetaxel treatment to crossover to receive JDQ443 treatment regardless of progression on docetaxel.

The study population will include adult participants with locally advanced or metastatic (stage IIIB/IIIC or IV) KRAS G12C mutant non-small cell lung cancer (by tissue or plasma as determined by a Novartis-designated central laboratory or accepted local tests) who have received prior platinum-based chemotherapy and prior immune checkpoint inhibitor therapy administered either in sequence or as combination therapy.

Approximately 360 participants will be randomized to JDQ443 or docetaxel in a 1:1 ratio stratified by prior line of therapy and ECOG performance status.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically confirmed locally advanced/metastatic (stage IIIB/IIIC or IV)
* Participant has a KRAS G12C mutation present in tumor tissue or plasma prior to enrollment, as determined by a Novartis designated central laboratory or by accepted local tests.
* Participants has received one prior platinum-based chemotherapy regimen and one prior immune checkpoint inhibitor therapy for locally advanced or metastatic disease
* Participant has at least 1 evaluable (measurable or non-measurable) lesion by RECIST 1.1 at the screening visit.

Exclusion Criteria:

* Participants who have previously received docetaxel (except if received in neoadjuvant or adjuvant setting with no progression within 12 months after the of end of treatment), or any other KRAS G12C inhibitor.
* Participant has EGFR-sensitizing mutation and/or ALK rearrangement by local laboratory testing. Participants with other druggable alterations will be excluded if required by local guidelines.
* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Participant has an history of interstitial lung disease or pneumonitis grade > 1.

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Approximately up to 24 months
  PFS is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is based on central assessment and using RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately up to 33 months
  OS is defined as the time from date of randomization to date of death due to any cause
Overall Response Rate (ORR) | Approximately up to 33 months
  ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) based on central and local investigator's assessment according to RECIST 1.1.
Disease Control Rate (DCR) | Approximately up to 33 months
  DCR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Non-CR/Non-PD.
Time To Response (TTR) | Approximately up to 33 months
  TTR is defined as the time from the date of randomization to the date of first documented response (CR or PR, which must be confirmed subsequently)
Duration of Response (DOR) | Approximately up to 33 months
  DOR is calculated as the time from the date of first documented response (complete response (CR) or partial response (PR)) to the first documented date of progression or death due to underlying cancer.
Progression-Free Survival after next line therapy (PFS2) | Approximately up to 33 months
  PFS2 (based on local investigator assessment) is defined as time from date of randomization to the first documented progression on next line therapy or death from any cause, whichever occurs first.
Concentration of JDQ443 and its metabolite in plasma | Approximately up to 33 months
  To characterize the pharmacokinetics of JDQ443 and its metabolite HZC320
Time to definitive deterioration of Eastern Cooperative Group of Oncology Group (ECOG) performance status | Approximately up to 33 months
  Deterioration of Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Time to definitive 10-point deterioration symptom scores of chest pain, cough and dyspnea per QLQ-LC13 | Approximately up to 33 months
  The EORTC QLQ LC13 is a 13-item, lung cancer specific questionnaire module, and it comprises both multi-item and single-item measures of lung cancer-associated symptoms (i.e. coughing, hemoptysis, dyspnea and pain) and side-effects from conventional chemo- and radiotherapy (i.e. hair loss, neuropathy, sore mouth and dysphagia). The time to definitive 10-point deterioration is defined as the time from the date of randomization to the date of event, which is defined as at least 10 points absolute increase from baseline (worsening), with no later change below the threshold or death due to any cause
Time to definitive 10-point deterioration in global health status/QoL, shortness of breath and pain per QLQ-C30 | Approximately up to 33 months
  The EORTC QLQ-C30 is a questionnaire developed to assess the health-related quality of life of cancer participants. The questionnaire contains 30 items and is composed of both multi-item scales and single-item measures based on the participants experience over the past week. These include five domains (physical, role, emotional, cognitive and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/HRQoL scale. The time to definitive 10-point deterioration is defined as the time from the date of randomization to the date of event, which is defined as at least 10 points absolute increase from baseline (worsening) of the corresponding scale score, with no later change below the threshold or death due to any cause
Change from baseline in EORTC-QLQ-C30 | Approximately up to 33 months
  The EORTC QLQ-C30 is a questionnaire developed to assess the health-related quality of life of cancer participants. The questionnaire contains 30 items and is composed of both multi-item scales and single-item measures based on the participants experience over the past week. These include five domains (physical, role, emotional, cognitive and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/HRQoL scale. A higher score indicates a higher presence of symptoms.
Change from baseline in EORTC-QLQ-LC13 | Approximately up to 33 months
  The EORTC QLQ LC13 is a 13-item, lung cancer specific questionnaire module, and it comprises both multi-item and single-item measures of lung cancer-associated symptoms (i.e. coughing, hemoptysis, dyspnea and pain) and side-effects from conventional chemo- and radiotherapy (i.e. hair loss, neuropathy, sore mouth and dysphagia). A higher score indicates a higher presence of symptoms.
Change from baseline in EORTC-EQ-5D-5L | Approximately up to 33 months
  The EQ-5D-5L is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression.
Change from baseline in NSCLC-SAQ | Approximately up to 33 months
  The Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) is a 7-item, patient-reported outcome measure which assess patient-reported symptoms associated with advanced NSCLC. It contains five domains and accompanying items that were identified as symptoms of NSCLC: cough (1 item), pain (2 items), dyspnea (1 item), fatigue (2 items), and appetite (1 item).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (52):
- Valley Medical Center Research, Renton, Washington, United States
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Pilar, Buenos Aires
- Australia (2):
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
- Canada (2):
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (9):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Chongqing
- Novartis Investigative Site, Turku, Finland
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion Crete.
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Reykjavik, Iceland
- India (2):
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Delhi
- Italy (3):
  - Novartis Investigative Site, Lucca, LU
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Amman, Jordan
- Novartis Investigative Site, Ed Daoura, Lebanon
- Malaysia (2):
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Novartis Investigative Site, Mexico City, Mexico
- Portugal (2):
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Cluj-Napoca, Cluj, Romania
- Novartis Investigative Site, Ljubljana, Slovenia
- Novartis Investigative Site, Seongnam-si, Gyeonggi-do, South Korea
- Spain (4):
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Tainan, Taiwan
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Adana, Adana
  - Novartis Investigative Site, Ankara, Bilkent-Cankaya
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Istanbul, Pendik
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Ankara
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.